CLINICAL TRIAL: NCT04723901
Title: Clinical Trial of CD19/CD22 Dual Target CAR-T Cells in the Treatment of Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: Dual Target CAR-T Cells in B-cell Acute Lymphoblastic Leukemia
Acronym: CAR-T
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-005
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Dual-target CAR-T Cells; B ALL; Relapse; Refractory B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Dual target CAR-T cell therapy
  Interventions: Biological: Dual target CAR-T cell therapy

INTERVENTIONS:
Biological: Dual target CAR-T cell therapy — CD19/CD22 dual target CAR-T cell therapy

SUMMARY:
Prospectively evaluate the safety and effectiveness of CD19/CD22 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Prospectively evaluate the safety and effectiveness of CD19/CD22 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell acute lymphoblastic leukemia. Strictly follow the inclusion criteria to screen eligible subjects for inclusion in clinical trials. The selected patients received CD19/CD22 dual-target CAR-T cell therapy. After the treatment is over, follow-up regularly to determine the survival status and follow-up treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to participate in this study:

  1. 14-75 years old, no gender limit;
  2. According to the 2020 World Health Organization (WHO) diagnostic criteria, it is diagnosed as relapsed/refractory B-cell acute lymphoblastic leukemia (r/r B-ALL);
  3. ECOG behavior status score is 0-2 points;
  4. Expected survival time ≥ 3 months;
  5. No contraindications to peripheral apheresis;
  6. Flow cytometry confirms that the original cells express CD22;
  7. Those who are tolerant to CD19 CAR-T cell therapy or those with low CD19 expression;
  8. No serious heart, lung, liver or kidney disease;
  9. Ability to understand and willing to sign the informed consent form for this trial.

Exclusion Criteria:

* Patients with any of the following cannot be included in this study:

  1. The original cells expressing CD19 and CD22 are negative;
  2. There is active infection;
  3. Abnormal liver function ( glutamic-pyruvic transaminase>1.5×ULN, glutamic oxalacetic transaminase>2.5×ULN), abnormal renal function (serum creatinine>1.5×ULN);
  4. People with unstable angina or New York Heart Association class 3/4 congestive heart failure, multiple organ dysfunction;
  5. HIV/AIDS patients;
  6. Those who need long-term anticoagulation (warfarin or heparin), antiplatelet (aspirin, dose>300mg/d; clopidogrel, dose>75mg/d) treatment;
  7. Those who received radiotherapy within 4 weeks before the start of the study (blood sampling);
  8. Known or suspected drug abuse or alcohol dependence;
  9. People with mental illness or other conditions cannot obtain informed consent, and cannot cooperate with the requirements for completing the experimental treatment and inspection procedures;
  10. Those who have participated in other clinical trials within 30 days;
  11. Pregnant or lactating women, male subjects (or their partners) or female subjects have a pregnancy plan during the study period to 6 months after the end of the test, and are unwilling to use a medically approved effective contraceptive measure during the test period (Such as intrauterine device or condom);
  12. The investigator judged that it is not suitable to participate in this trial.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | From date of initial treatment to the end of follow up, up to 2 years
  1. No blasts in peripheral blood, no extramedullary leukemia;
  2. Three-line bone marrow hematopoietic recovery, primitive cells <5%;
  3. Peripheral blood absolute neutrophil count>1.0×10^9/L;
  4. Peripheral blood platelet count>100×10^9/L;
  5. No recurrence within 4 weeks

SECONDARY OUTCOMES:
Overall survival rate | From admission to the end of follow up, up to 2 years.
  The proportion of surviving patients at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
no intention